CLINICAL TRIAL: NCT05130593
Title: Pilot Study Evaluating the Hedonic Acceptability and Absorption of the Bioactive Compounds of a 5011-Nutrasorb Bar (Russian Tarragon Nutrasorb)
Brief Title: Pilot Study Evaluating the Acceptability and Absorption of the Bioactive Compounds of a Russian Tarragon Nutrasorb Bar
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Jennifer C. Rood, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2020-022; 5P50AT002776-15 (NIH)
Record Dates: First submitted 2021-10-06; First posted 2021-11-23 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Prevention
Keywords: tarragon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nutrasorb bar evaluation: Participants in Phase 1 will taste test the bar for acceptability. Participants in Phase 2 will consume the bar and have blood samples drawn for measurement of safety parameters (glucose and insulin) and bioactive compounds (DMC-2).
  Interventions: Dietary Supplement: Nutrasorb bar

INTERVENTIONS:
Dietary Supplement: Nutrasorb bar — 250 kcal bar containing 30 g of 5011-Nutrasorb (120 kcal), 20 g fat (100 kcal), and 30 kcal from carbohydrate and flavorings

SUMMARY:
The purpose of this study is to make a bar from the soy-protein Russian Tarragon complex (PMI-5011/Nutrasorb) that is safe and acceptable for consumption, and to test the blood levels of plasma bioactive (DMC-2) after ingestion of the bar. The PMI-5011/Nutrasorb comes from a plant source called Artemisia dracunculus. This plant has a long history of medicinal (health) and culinary (food) use and has been reported as effective as a traditional treatment for diabetes in various parts of the world.

DETAILED DESCRIPTION:
Phase 1

Test Day: Fasting Visit (nothing to eat or drink other than water beginning at 10 pm the night before the test day); visit will be approximately 1 ½ hours.

The following procedures will be done on the Test Day:

* Informed consent will be signed by those agreeing to participate.
* Body weight and height will be measured (body mass index will be calculated from these measures).
* Participants will provide a list of any medications they are currently taking.
* Blood pressure and pulse will be measured.
* Taste test of the study bar will be conducted.
* Participants will answer questions regarding the appearance, smell, taste, texture, aftertaste, and pleasantness of the bar.

Phase 1 participants may be asked to return up to two additional times to complete the taste test and questions again. This will occur if the product is found unacceptable and will be completed after a new bar is produced.

Phase 2

Screening Visit: Fasting Visit (nothing to eat or drink other than water after 10 pm the night before the Screening Visit); visit will be approximately 1 ½ hours.

The following procedures will be done on the Screening Visit:

* Informed consent will be signed by those agreeing to participate.
* Body weight and height will be measured (body mass index will be calculated from these measures).
* Blood pressure and pulse will be measured.
* Medical history questionnaire will be completed.
* Blood will be drawn (approximately 2 teaspoons) to assess overall health.

Test Day: Fasting visit (nothing to eat or drink other than water after 10 pm the night before the Test Day); visit will be approximately 4 hours and will be completed within 30 days after Screening Visit.

The following procedures will be done on the Test Day:

* Blood will be drawn from an IV line placed in the participant's arm to assess the level of nutrients, blood sugar levels, and insulin levels from the study bar 10 minutes before the bar is consumed, immediately after the bar is consumed, and 30, 60, 120, and 180 minutes after the bar is consumed. A total of approximately 6 teaspoons of blood will be drawn for this Test Day.
* Participants will answer questions regarding the appearance, smell, taste, texture, aftertaste, and pleasantness of the bar.
* Participants will be asked about any side effects and how they feel throughout the Test Day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females between 18 and 50 years of age inclusive.
* Body mass index between 20-30 kg/m2.

Exclusion Criteria:

* Pregnant or currently lactating.
* Taking any prescription medications.
* Taking any over-the-counter medications that cannot be stopped for test days.
* Allergic to any ingredients contained in the bar.
* Other conditions or situations that would interfere with the study or the participant's safety as determined by the investigators.
* Participants in Phase 1 of the study may not participate in Phase 2 of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy males and females aged 18-50 with a body mass index between 20-30 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Rood, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Participants taste-tested a bar containing PMI-5011/Nutrasorb for acceptability. Nutrasorb bar: 250 kcal bar containing 30 g of 5011-Nutrasorb (120 kcal), 20 g fat (100 kcal), and 30 kcal from carbohydrate and flavorings
- Phase 2: Participants consumed a bar containing PMI-5011/Nutrasorb and had blood samples drawn for measurement of safety parameters (glucose and insulin) and bioactive compounds (DMC-2). Nutrasorb bar: 250 kcal bar containing 30 g of 5011-Nutrasorb (120 kcal), 20 g fat (100 kcal), and 30 kcal from carbohydrate and flavorings
Period: Overall Study
Arm/Group | Phase 1 | Phase 2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 7 | 10 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Palatability of Bar
Description: Participants were asked to rate the bar on a visual analog scale to indicate their impression of its visual appearance, smell, taste, texture, aftertaste, and overall pleasantness. The scale range for each attribute is 0-100 with higher scores equating to a better outcome.
Time Frame: Test Day (immediately after taste-testing the bar)
Population: Only the participants in Phase 1 of the study participated in taste-testing of the bar for palatability. Participants from Phase 1 were not allowed to participate in Phase 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1
Number analyzed (Participants) | 10
score on a scale
  Visual Appearance | 77.4 (19.7)
  Smell | 59.5 (19.2)
  Taste | 27.8 (24.4)
  Texture | 50.6 (20.8)
  Aftertaste | 56.5 (31.4)
  Pleasantness | 32.2 (25.6)

2. Secondary Outcome: Levels of Plasma BIoactive (DMC-2) Before and After Ingestion of a Bar Containing PMI-5011/Nutrasorb.
Description: Participants consumed a bar containing PMI-5011 and Nutrasorb and had blood samples drawn for measurement of DMC-2. Nutrasorb bar: 250 kcal bar containing 30 g of PMI-5011/Nutrasorb (120 kcal), 20 g fat (100 kcal), and 30 kcal from carbohydrate and flavorings
Time Frame: 10 minutes pre-consumption, immediately post-consumption, and 30, 60, 120, and 180 minutes post-consumption
Population: Only the participants in Phase 2 of the study had blood samples drawn for measurement of bioactive compounds (DMC-2). Participants from Phase 1 were not allowed to participate in Phase 2.
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Phase 2: Participants consumed a Nutrasorb bar and had blood samples drawn for measurement of safety parameters (glucose and insulin) and bioactive compounds (DMC-2). Nutrasorb bar: 250 kcal bar containing 30 g of 5011-Nutrasorb (120 kcal), 20 g fat (100 kcal), and 30 kcal from carbohydrate and flavorings
Arm/Group | Phase 2
Number analyzed (Participants) | 10
ug/mL
  - 10 min | 0.05 (0.00)
  0 min | 0.05 (0.00)
  30 min | 0.094 (0.026)
  60 min | 0.076 (0.022)
  120 min | 0.087 (0.026)
  180 min | 0.074 (0.013)

3. Secondary Outcome: Levels of Serum Glucose Before and After Ingestion of a Bar Containing PMI-5011/Nutrasorb.
Description: Participants consumed a bar containing PMI-5011 and Nutrasorb and had blood samples drawn for measurement of safety parameters (glucose). Nutrasorb bar: 250 kcal bar containing 30 g of 5011-Nutrasorb (120 kcal), 20 g fat (100 kcal), and 30 kcal from carbohydrate and flavorings
Time Frame: 10 minutes pre-consumption, immediately post-consumption, and 30, 60, 120, and 180 minutes post-consumption
Population: Only the participants in Phase 2 of the study had blood samples drawn for measurement of serum glucose. Participants from Phase 1 were not allowed to participate in Phase 2.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Phase 2
Number analyzed (Participants) | 10
mg/dL
  -10 min | 88 (6.2)
  0 min | 89 (5.5)
  30 min | 91 (6.9)
  60 min | 91 (5.5)
  120 min | 90 (4.7)
  180 min | 89 (5.1)

4. Secondary Outcome: Measurement of Blood Levels of Serum Insulin Before and After Ingestion of a Bar Containing PMI-5011/Nutrasorb.
Description: Participants consumed a bar containing PMI-5011 and Nutrasorb and had blood samples drawn for measurement of safety parameters (insulin). Nutrasorb bar: 250 kcal bar containing 30 g of 5011-Nutrasorb (120 kcal), 20 g fat (100 kcal), and 30 kcal from carbohydrate and flavorings
Time Frame: 10 minutes pre-consumption, immediately post-consumption, and 30, 60, 120, and 180 minutes post-consumption
Population: Only the participants in Phase 2 of the study had blood samples drawn for measurement of insulin. Participants from Phase 1 were not allowed to participate in Phase 2.
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Phase 2
Number analyzed (Participants) | 10
uIU/mL
  -10 min | 9.6 (12.8)
  0 min | 10.4 (13.9)
  30 min | 30.7 (30.5)
  60 min | 25.8 (31.4)
  120 min | 14.3 (16.7)
  180 min | 7.2 (6.4)

ADVERSE EVENTS:
Time Frame: Test Day (up to 4 hours)
Arm/Group | Phase 1 | Phase 2
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT05130593/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT05130593/ICF_001.pdf